CLINICAL TRIAL: NCT04186689
Title: Relationship Between Food Insecurity, Maternal Psychological Status, and Child Dental Behavior: a Cross-Sectional Study
Brief Title: Relationship Between Food Insecurity and Child Dental Anxiety
Acronym: FI
Status: Completed | Type: Observational
Sponsor: dina darwish (Other)
Responsible Party: Sponsor-Investigator, dina darwish, principle investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: 829
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Food Insecurity; Child Dental Anxiety; Maternal Psychological Distress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- children in fully food secure households (G1): preschool children live in a fully food secure household have at least a carious tooth that needs treatment under local anesthesia other than extraction without any previous dental treatment experience.
  Interventions: Other: Routine Dental Examination
- children in marginally food secure households (G2): preschool children live in a marginally food secure household have at least a carious tooth that needs treatment under local anesthesia other than extraction without any previous dental treatment experience.
  Interventions: Other: Routine Dental Examination
- children in food insecure households (G3): preschool children live in a food-insecure household have at least a carious tooth that needs treatment under local anesthesia other than extraction without any previous dental treatment experience.
  Interventions: Other: Routine Dental Examination

INTERVENTIONS:
Other: Routine Dental Examination — Routine dental examination for the pre-school children Questionnaire for their mothers

SUMMARY:
identifying children with dental anxiety among those who suffered from food insecurity will enable to implement preventive strategies and early intervention. The aim of this study is to examine the relationship between food insecurity, maternal psychological status and child dental behavior.

DETAILED DESCRIPTION:
A well-trained investigator will collect data on maternal age (in years), the marital status, the educational levels of both parents and their employment status, pregnancy information, as well as family structure (whether children are living with both parents or not), number of siblings (none, one, two, or ≥three). Information on family monthly income and crowding index which is defined as the average number of people per room, excluding both the kitchen and bathrooms will be also obtained.

The level of household food insecurity will be determined using the validated Arabic version of the Household Food Insecurity Access Scale (HFIAS) which categorizes food insecurity into three levels (food secure , marginally food secure and food insecure) where the final score is given according to the sum of affirmative responses to the tool statements and the higher the score the more the level of food insecurity.

The validated Arabic version of the 14-item Perceived Stress Scale will be used to measure the self-reported level of stress among mothers of the enrolled children by assessing their feelings and thoughts during the last month. The level of child's dental anxiety will be assessed during the initial oral examination before starting any dental treatment procedures using the six-point Venham behavior rating scale which ranges from total cooperation (0) to no cooperation

ELIGIBILITY:
Inclusion Criteria:

* the selected children accompanied by their mother should fulfill the following inclusion criteria:

  * Age range 3.5-6 years
  * Having at least one tooth with dental caries indicated for dental treatment under local anesthesia other than extraction
  * Visiting the dental clinic for the first time

Exclusion Criteria:

* Children with the following criteria will be totally excluded from the study: Have any medical/neurological, communicative or developmental disorders as well as children with special healthcare needs.

Ages: 40 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: study populations are healthy pre-school children( 3.5-6 years old)having at least one tooth needs dental treatment, accompanied by their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
A six-point Venham Behavior Rating Scale to evaluate the child behavior during dental examination scale score from(0)the best outcome to (6) worst outcome | 6 months
  which ranges from total cooperation (0) to no cooperation(6)
questionnaire containing 2 scales Household Food Insecurity Access Scale( score food secure better outcome -severely food insecure the worst outcome) and 14-item Perceived Stress Scale (scores from 0 better outcome to 40 worst outcome) | 6 months
  to measure the effect of the predictor variable and the potential mediators which are the household food insecurity and maternal psychological status respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Dina D Abd-Elmoneam, masters, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the exact plan to share individual participant data (IPD) is still not formulated, once it is ready I will share.